CLINICAL TRIAL: NCT00283647
Title: MR Assessment of Brain Function Altered by Lead Exposure
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 11261-CP-004
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Lead Exposure
Keywords: lead exposure; magnetic resonance imaging; magnetic resonance spectroscopy; functional magnetic resonance; brain development

SUMMARY:
Exposure to lead during pregnancy, infancy, and childhood increases the individual likelihood of impaired school performance, increased impulsiveness, aggression, and delinquent behavior. Disorders that result from exposure to environmental neurotoxicants are a complex web of interactions between genetic, neurochemical, biochemical, environmental and social factors that influence children during critical periods of development. To date, research in the area of human developmental neurotoxicology focuses primarily on global measures of sensory-motor development and cognition. However, studies elucidating the biological basis for developmental and behavioral disorders due to environmental toxicant exposure are lacking. Although gross brain structure appears normal, underlying problems exist at a neural level. Our proposal seeks to relate childhood environmental lead exposure at various levels and stages of development with detriments in brain structure and neurochemical functioning assessed with magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). Cortical and subcortical brain volumes will be determined with high resolution MRI. Neuronal and glial cell markers will be measured using proton MRS. These structural and chemical measures will also be correlated with behavioral measures from the young adult participants of the Cincinnati Lead Study (CLS). These participants represent a unique and ideal cohort of approximately 240 subjects with detailed histories of exposure and behavioral outcomes in lead exposed children monitored for approximately 20 years. A pilot study examining language, working memory and attention in combination with functional magnetic resonance imaging (fMRI) will also be performed to better understand the functional and behavioral deficits.

DETAILED DESCRIPTION:
Overview of Imaging

All MRI and MRS investigations will be acquired on a 1.5 clinical MR scanner. The MRI and MRS procedures will take approximately a half-hour to complete. Subjects also having fMRI performed will require another scanning session on the research 3T MR scanner with one hour for completion. Orientation to the scanning procedures will take place during the visit to the Imaging Research Center, upon completion of informed consent. The subject will be given a brief introduction to the general MR scanning procedures and demonstration of the MRI machinery. Prior to beginning studies, subjects will be allowed to familiarize themselves with the scanner to decrease anxiety about the experiment. Subjects will receive instruction and practice in the appropriate behaviors necessary for a successful MR study. The research MR technologist has over 10 years experience in pediatric neuroimaging and takes great care to make subjects comfortable in the head coil so that they can remain as motionless as possible for the duration of the scan. The subject is asked to select a video to watch and is given the video goggles to focus and adjust to fit, immediately upon entering the scanner room. Once on the table, the subject's head is restrained within a padded head holder with additional foam pads, while the subject is watching the video. This arrangement is snug but not uncomfortable. The subject is asked to hold a button box in one hand; this will be used to make responses that will provide performance data used for validity checks on task engagement as well as correlation with the activation results. A "panic ball" will also be provided to each subject. The subjects will be carefully oriented to the equipment and environment and will engage in explicit practice of all of the task requirements.

Anatomical Localizer and High Resolution Imaging Acquisitions

After subjects are positioned in the scanner, the scanner will be shimmed to provide a homogeneous magnetic field for image acquisition. An initial alignment scan is done in 3 orthogonal planes simultaneously using a fast gradient echo sequence developed for the scanner. This scan takes approximately 30 seconds and provides a quick view of the subject's head position. Next, a high-resolution T1-weighted 3-D neuroanatomic scan will be obtained using a inversion recovery, fast spoiled gradient echo (IR-prepped FSPGR) protocol to provide images for morphometric studies, localization of MRS and anatomical localization of the activation maps. The acquisition takes approximately 6 minutes and yields a minimum spatial resolution of 1mm x 1mm x 1.5mm with sufficient signal to noise ratio and contrast between gray and white matter for both manual and semi-automated segmentation of regional brain volumes.

Proton MR Spectroscopy Acquisitions

Proton MR spectroscopy data is acquired using the point resolved spectroscopy localization (PRESS) method. Graphically, 3D cubic volume elements "voxels" are positioned in the anatomic locations based upon the 3D images. Voxel 1 is placed in the anterior cingulate, voxel 2 the left dorsalateral prefrontal cortex, voxel 3 within the basal ganglia encompassing the caudate, putamen and internal capsule and voxel 4 is placed along the superior temporal gyrus. Voxel 5 is used as a control and is positioned in the left centrum semiovale, a believed to be unaffected white matter region. Voxels 6 and 7 are positioned within the cerebellum and vermis, respectively.

Functional MRI Acquisitions

The location of the 24 axial slices to be imaged in the fMRI procedures is identified from the high resolution anatomical imaging sequence. These 24 slices, 5 millimeters thick (120 mm), are sufficient to cover areas extending superiorly from below the inferior aspect of the cerebellum to the apex of the cerebrum in an adult brain. Subjects undergo the fMRI scan sequence during which they will be asked to perform tasks which can involve language, memory and attention. The protocol for the fMRI scans will be a T2 - weighted gradient -echo Echo Planar Imaging (EPI) method. The time sequence of alternating periods (30 sec) of task conditions is repeated 5.5 times for a total of 11 intervals with 10 acquisitions per interval, resulting in 240 images. 24 image slices are acquired for each time point. Synchronization of the fMRI scans with the video stimuli is fully automated so that when the visual presentation commences on the Macintosh computer, it triggers the Bruker MR scanner to begin acquisitions. The MacStim presentation and the fMRI scan timing are synchronized from the trigger point to the end of the experiment. The high resolution MDEFT sequence allows for the 24 fMRI scan planes to be extracted from this 3D anatomical data set by interpolation for use as an anatomical underlay for the activation maps.

Testing paradigms

The Verb Generation task is based on that described by Binder et al. and involves the auditory presentation of a series of nouns. The subject is required to generate verbs that are associated with each noun. For example, if the noun "ball" is presented, the subject might generate the verbs "throw," "kick," and "hit." The subject is instructed to think the verbs silently, without saying them, in order to minimize the motion artifact associated with speech. Task performance is monitored by a button push each time the subject thinks of a verb. This expressive task is assumed to require the engagement of dominant frontal lobe and parietal lobe language areas. This task is derived from the clinical literature as an MRI analog of the procedure used in the Wada test. It is now widely used for testing hemispheric dominance for language in adults. It is included in the current protocol partly to provide a point of comparison with the existing literature as well as with our own preliminary data from other populations. Finally, this is a difficult semantic task and fits neatly into the scope of the language skills we are seeking to monitor with lead exposed young adults.

For studies designed to examine working memory, the "n-back" tasks are administered using MacStim software on a Macintosh PowerBook laptop computer. The "n-back" is a working memory task in which subjects view numbers from one to four that consistently appear in one of four quadrants on the screen. Subjects view the stimuli through the audiovisual goggle system and respond using a button box on which the buttons had been arranged so as to correspond with the numbers appearing on the screen. In the "zero back" condition, subjects press the number that corresponds to the number then appearing. In the "two back" condition, the subject presses the button corresponding to the number that appeared two places prior to the number then on the screen. During the fMRI scans, subjects are asked to perform the "zero and two back" tasks in a block-periodic design. During each condition, 15 numbers appear over a 30 second interval. In all, 11 intervals are presented over a 5 1/2 minute scan. The "zero-back" task serves as the contrast for the "two back" tasks. Data from the first "zero back" task interval is discarded during post-processing to avoid any non-equilibrium intensity modulation effects.

In assessing attention, the CPT-IP is administered using MacStim software and MRI compatible audiovisual system. During the fMRI scans subjects are asked to perform the CPT-IP task in a block-periodic design. Participants alternate between two conditions. During the first condition, subjects perform in a control task during which they view a four-digit number repeating at a constant rate (0.75 sec.) and are instructed to simply look at the flashing number without responding in any way. During the second condition, subjects watch a series of high resolution four digit numbers appearing in a random sequence and are instructed to press a response button when they see any number repeat twice in a row during the sequence. Numbers again appear every 0.75 sec.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in the Cincinnati Lead Study.
2. Age range of at least 18 years with an upper limit of 25 years.
3. Negative history for metabolic, neurologic, cardiac disease.
4. Negative family history for metabolic or neurologic disease (in first-degree relatives only) to include genetic disorders.

Exclusion Criteria:

1. Presence of an implant such as a hearing aid, cochlear implant, pacemaker or neuro-stimulator containing electrical circuitry or generating electrical signals or having moving metal parts.
2. Presence of metal implants, orthopedic pins or plates above the level of the waist.
3. Presence of orthodontic braces.
4. Subjects who demonstrate or express noticeable anxiety and/or cannot readily communicate with personnel operating the MR equipment will be excluded.
5. Pregnancy.

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2002-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Cecil, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Dept. of Radiology and the Imaging Research Center, Cincinnati, Ohio, United States